CLINICAL TRIAL: NCT04541745
Title: Prospective Cohort Study Comparing Functional Recovery Following Orthopedic Wrist Surgery Under Peripheral Nerve Block Versus General Anesthesia
Brief Title: Functional Recovery Following Orthopedic Wrist Surgery Under Peripheral Nerve Block Versus General Anesthesia
Acronym: FUNCTION
Status: Completed | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Jennifer Héroux, Anesthesiology and CIP resident, Université de Sherbrooke
Other Study IDs: 2020-3241
Record Dates: First submitted 2020-07-29; First posted 2020-09-09 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Recovery of Function
Keywords: Upper limb surgery; Functional recovery; Postoperative recovery; General anesthesia; Brachial plexus; Nerve block; Regional anesthesia; Peripheral anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims at determining if there is an association between locoregional anesthesia and postoperative functional recovery for orthopedic surgery to repair a distal radial fracture, as compared to general anesthesia.

DETAILED DESCRIPTION:
All patients undergoing orthopedic wrist surgery under locoregional or general anesthesia at the CIUSSS de l'Estrie-CHUS who meet the selection criteria will be approach to participate in this prospective single-center observational study. Using the visual analog scale and anesthesia scale, the pain and the satisfaction of the patient will be evaluated respectively 2 weeks postoperatively. At the second visit, 6 to 8 weeks postoperatively, the participant will complete the QuickDASH questionnaire to evaluate his functional recovery and the participant's pain will be reassessed with the visual analogue scale. Finally, 12 weeks postoperatively, the wrist-joint range of motion and grip-strength test results will be recorded. The participant will also be asked to complete the QuickDASH and PRWE (Patient-Rated Wrist Evaluation) questionnaires to reevaluate his functional recovery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and more
* American Society of Anesthesiologists (ASA) score I, II, or III
* Single distal radial fracture with or without ulna involvement
* Orthopedic surgery by open reduction of the wrist for a distal radial fracture with or without ulnar involvement

Exclusion Criteria:

* Active pregnancy
* Surgery with combined anesthesia (locoregional and general)
* Locoregional anesthesia with catheter insertion for postoperative analgesia
* Individuals with chronic pain as defined by preexisting neuropathy of the operated arm, preexisting radiculopathy of the operated limb, complex regional pain syndrome, or fibromyalgia
* Polytrauma
* Inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patient cohort will be composed of all patients undergoing orthopedic wrist surgery under locoregional or general anesthesia at the CIUSSS de l'Estrie-CHUS who meet the selection criteria.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Functional recovery using the QuickDASH (Quick Disabilities of Arm, Shoulder and Hand) questionnaire | 12 weeks post-surgery
  The QuickDASH assess the functional recovery. It consists of 11 questions scored from 1 to 5 (1 = no difficulty to 5 = unable). Higher scores indicate a greater level of disability.
Functional recovery using the PRWE (Patient Rated Wrist Evaluation) Questionnaire | 12 weeks post-surgery
  The PRWE (Patient Rated Wrist Evaluation) Questionnaire assess the pain and the persistence of functional difficulty in activities of daily living following wrist surgery. It consists of 15 questions, each rated on a scale from 0 to 10. Five questions deal specifically with pain and are rated as 0 (no pain) to 10 (worse pain); 10 questions are on functional recovery, rated from 0 (no difficulty) to 10 (unable to do). Higher scores on the subscales represent greater pain or functional disability.
Functional recovery using the range of motion of all movement of the wrist | 12 weeks post-surgery
  We evaluate the range of motion of all movement of the wrist with a goniometer
Functional recovery using the grip strenght | 12 weeks post-surgery
  We evaluate the grip strength with JAMAR hydraulic hand dynamometer. The participant squeezes the device as hard as they can. We averaged three values on both sides.

SECONDARY OUTCOMES:
Pain- 2 weeks | 2 weeks post-operative
  Post-operative pain score on the visual analogue scale. It is a 10 cm line on which the patient indicate their level of pain between 0 cm (no pain) and 10 cm (worst pain of their life).
Pain - 6 weeks | 6 weeks post-operative
  Post-operative pain score on the visual analogue scale. It is a 10 cm line on which the patient indicate their level of pain between 0 cm (no pain) and 10 cm (worst pain of their life).
Functional recovery at 6 weeks | 6 weeks post-operative
  Functional recovery following an orthopedic surgery under peripheral nerve block versus general anesthesia using the QuickDASH (The Quick Disabilities of Arm, Shoulder and Hand). The questionnaire consists of 11 questions scored from 1 to 5 (1 = no difficulty to 5 = unable). When all the questions are answered, the questionnaire calculate a percentage of disability. Higher scores indicate a greater level of disability.
Patient satisfaction | 2 weeks post-operative
  Satisfaction score on the visual analogue scale. It is a 10 cm line on which the patient indicate their level of satisfaction between 0 cm (not satisfied) and 10 (fully satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Frédérick D'Aragon, Study Director — Université de Sherbooke
Locations (1):
- CIUSSS de l'estrie- CHUS, Sherbrooke, Quebec, Canada

REFERENCES:
- [Derived] Heroux J, Bessette PO, Bedard S, Lamarche D, Gagnon A, Echave P, Loignon MJ, Patenaude N, Baillargeon JP, D'Aragon F. Functional recovery of wrist surgery with regional versus general anesthesia: a prospective observational study. Can J Anaesth. 2024 Jun;71(6):761-772. doi: 10.1007/s12630-023-02615-y. Epub 2023 Nov 6. PMID 37932649
- [Derived] Heroux J, Bessette PO, Belley-Cote E, Lamarche D, Echave P, Loignon MJ, Patenaude N, Baillargeon JP, D'Aragon F. Functional recovery with peripheral nerve block versus general anesthesia for upper limb surgery: a systematic review. BMC Anesthesiol. 2023 Mar 24;23(1):91. doi: 10.1186/s12871-023-02038-8. PMID 36964490